CLINICAL TRIAL: NCT01354158
Title: A Dose Response Trial of Droxidopa to Treat Hypotension in Persons With SCI
Brief Title: A Dose Titration of Droxidopa in Patients With Spinal Cord Injury
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bronx VA Medical Center (U.S. Federal Agency)
Collaborators: Chelsea Therapeutics (Industry)
Responsible Party: Jill M. Wecht/Health Science Specialist, James J. Peters VA Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01272
Record Dates: First submitted 2011-05-12; First posted 2011-05-16 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2011-05

CONDITIONS: Spinal Cord Injury; Hypotension
MeSH Terms: conditions — Spinal Cord Injuries; Hypotension | interventions — Droxidopa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Droxidopa (Experimental): The dose-titration response to ascending doses of Droxidopa (placebo, 100mg, 200mg, 400mg) will be measured four separate days.
  Interventions: Drug: Droxidopa

INTERVENTIONS:
Drug: Droxidopa — Dose titration of placebo, 100mg, 200mg, 400mg of Droxidopa will be given to assess the effects of Droxidopa on blood pressure and cerebral blood flow.
  Other Names: L-DOPs

SUMMARY:
The investigators seek to determine the efficacy, duration of action and safety of escalating dose of droxidopa on systemic blood pressure, cerebral blood flow and vasoactive hormones and catecholamines during upright seated posture.

Primary Question:

1. What is the lowest dose of droxidopa that increases seated SBP to 115±5 mmHg in men and 105±5 mmHg in women?

* When does the defined increase in SBP occur after oral ingestion of droxidopa?
* How long does this dose of droxidopa sustain SBP at these levels?
* What are the vital signs and the subjective symptomology following droxidopa administration?

Secondary Question:

1. What is the MFV response to droxidopa administration in hypotensive individuals with SCI?

* Does an increase in SBP correspond to an increase in MCA MFV?

Tertiary Question:

1. What is the vasoactive hormone and catecholamine response to droxidopa administration in hypotensive individuals with SCI?

* Does droxidopa administration result in a change in APR, Aldo or NE in hypotensive individuals with SCI?

DETAILED DESCRIPTION:
Persons with spinal cord injury (SCI), due to partial to complete interruption of sympathetic pathways from the brainstem to the cardiovascular system are prone to blood pressure dysregulation including hypotension which is worsened during orthostasis. It is well established that orthostatic hypotension (OH) hinders the rehabilitation process during the acute phase of SCI but also may hamper the resumption of independence and activity in persons with chronic SCI. Surprisingly, only a few reports exist on the use and efficacy of an alpha receptor agonist (midodrine hydrochloride) to restore blood pressure to more normal levels in persons with tetraplegia. Our group has recently reported normalization of supine blood pressure with a relatively low dose of the nitric oxide synthase inhibitor (NOSi), nitro-L-arginine methyl ester (L-NAME). In addition to an alpha agonist and a NOSi, the use of a norepinephrine (NE) precursor, droxidopa, may be safe and efficacious for the treatment of orthostatic hypotension in a human model of SCI.

It has been demonstrated that the blood pressure-raising effect of 3,4-threo-dihydroxyphenylserine (droxidopa) occurs independently of the central nervous system in human models of neurologic OH by conversion to norepinephrine (NE) in neuronal and non-neuronal tissue. Oral droxidopa is taken up by the more peripheral sympathetic neurons, converted to NE, stored and released appropriately during postural stress. Droxidopa has been used for the effective treatment of OH in several human models of neurologically caused autonomic disorders, such as familial amyloid polyneuropathy, autoimmune autonomic neuropathy, pure autonomic failure, and multiple system atrophy . The effectiveness of droxidopa at improving orthostatic blood pressure in persons with SCI has not been studied. To date, only a single case on the use of the drug in a person with SCI has been reported and the use droxidopa in that case was successful. The purpose of this proposal is to determine the dose effectiveness, duration of action and any adverse events following droxidopa administration in hypotensive individuals with SCI.

To determine the efficacy, duration of action and safety of escalating dose of droxidopa on systemic blood pressure, cerebral blood flow and vasoactive hormones and catecholamines during upright seated posture.

Primary Question:

1. What is the lowest dose of droxidopa that increases seated SBP to 115±5 mmHg in men and 105±5 mmHg in women?

* When does the defined increase in SBP occur after oral ingestion of droxidopa?
* How long does this dose of droxidopa sustain SBP at these levels?
* What are the vital signs and the subjective symptomology following droxidopa administration?

Secondary Question:

1. What is the MFV response to droxidopa administration in hypotensive individuals with SCI?

* Does an increase in SBP correspond to an increase in MCA MFV?

Tertiary Question:

1. What is the vasoactive hormone and catecholamine response to droxidopa administration in hypotensive individuals with SCI?

* Does droxidopa administration result in a change in APR, Aldo or NE in hypotensive individuals with SCI?

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18 and 65,
* diagnosed with hypotension as defined above,
* able to provide informed consent

Exclusion Criteria:

* Known or suspected sensitivity to study medication or any of its ingredients,
* current smoker,
* known coronary heart and/or artery disease,
* hypertension,
* diabetes mellitus or insipidus,
* thyroid disease,
* closed angle glaucoma,
* acute illness,
* major surgery in the last 30 days,
* renal diseases,
* pregnancy,
* recent history (within the past year) of cocaine use,
* tricyclic antidepressants, monoamine oxidase inhibitors, and catechol-O-methyltransferase inhibitors,
* currently taking vasoconstricting medicines, such as Midodrine, ephedrine, dihydroergotamine, and the triptan class of migraine drugs,
* Use of a halogen based anesthetic such as Halothane in the past 12 hours
* Currently taking Isoproterenol and other catecholamine preparations
* Peripheral Arterial Disease,
* Abdominal Aortic Aneurysm,
* Cerebrovascular Disease (Including prior CVA or TIA),
* History of or active Congestive Heart Failure,
* Known Systolic Dysfunction

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-05; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
The lowest dose of droxidopa that increases seated SBP to 115±5 mmHg in men and 105±5 mmHg in women | 4 days
  4 day titration of Droxidopa (placebo day 1, 100mg day 2, 200mg day 3, 400mg day). Blood pressure will be collected at the arm and finger (photoplethysmography) in 15 minute intervals during the duration of the protocol (approximately six hours). The subject will also wear a 24 hour portable arm blood pressure cuff, to assess the effect of Droxidopa on blood pressure 24 hrs post intervention.

SECONDARY OUTCOMES:
The MFV response to droxidopa administration in hypotensive individuals with SCI | 4 days
  MFV will be measured each day at distinct time points to track cerebral blood flow during Droxidopa administration.
To assess the vasoactive hormone and catecholamine response to droxidopa administration in hypotensive individuals with SCI | 4 days
  The catecholamine response to Droxidopa will be measured a total of 6 times throughout each study day by antecubital venipuncture.

CONTACTS AND LOCATIONS:
Overall Officials: Jill M Wecht, EdD, Principal Investigator — James J. Peters VA Medical Center
Locations (1):
- James J. Peters VA Medical Center, The Bronx, New York, United States